CLINICAL TRIAL: NCT03059914
Title: A Histomorphometric Analysis of New Bone Formation Following Sinus Augmentation Using Two Different Bone Graft Materials. A Pilot Study in Humans.
Brief Title: A Histomorphometric Analysis Following Sinus Augmentation Using Two Different Bone Graft Materials.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Jaime Lozada, Professor Program Director Implant Dentistry, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5170069
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Missing Teeth
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- InterOss (Experimental): Maxillary sinus augmentation using ABBM Inteross ( Xenograft)
  Interventions: Device: InterOss
- Bio-oss (Active Comparator): Maxillary sinus augmentation using ABBM Bio-oss ( Xenograft)
  Interventions: Device: Bio-oss

INTERVENTIONS:
Device: InterOss — Anorganic bovine bone mineral - Xenograft
  Arms: InterOss
Device: Bio-oss — Anorganic bovine bone mineral ( Xenograft)
  Arms: Bio-oss

SUMMARY:
The purpose of this investigator-initiated study is to compare new bone formation through histomorphometric analysis following maxillary sinus augmentation using two different bone graft materials. A total of twenty, sinus augmentation via a lateral approach will be performed for subjects requiring sinus augmentation for implant placement and randomly divided into 2 groups. These subjects will receive one of two different bone graft materials: 1) Anorganic bovine bone matrix- InterOss (Group A), 2) Anorganic bovine bone matrix- Bio-oss (Group B). At the time of implant placement (eight months after the sinus augmentation procedure), two bone biopsies will be collected from augmented site for the histomorphometric analysis. The percentage of vital bone will be measured and analyzed statistically, also the following will be measured: percentage of non-vital bone, percentage of non-bone material , and the percentage of connective tissue.

DETAILED DESCRIPTION:
Bovine xenograft has been established as a gold standard in maxillary sinus floor augmentation. This study was initiated to compare two different types of bovine xenografts following maxillary sinus floor augmentation. The comparison will performed using histomorphometric analysis of bone cores removed from the grafted sites. The patients that meet the guidelines for maxillary sinus floor augmentation via lateral window approach are randomly assigned into control and test groups. The surgery is performed by the same surgeon under the same protocols. The subjects in Group A - test group receive InterOss bone graft and subjects in Group B- Control Group receive BioOss bone graft. After eight months of healing at the sites, the patients are subjected to CBCT evaluation in preparation for implant placement. At the time of implant placement the two bone cores are collected from each grafted site using trephine burs. One bone core is collected from the crestal bone that will be site of implant placement and the second bone core is collected from the lateral window area not to interfere with the implant site. These bone cores are stored intact inside the trephine burs, fixed, stored and transported to the lab for histomorphometric analysis. The following parameters are measured and reported after the histomorphometric analysis.

percentage of vital bone percentage of non-vital bone ( graft material) percentage of non-bone material percentage of connective tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old who are able to read and sign an informed consent form.
2. Patient who has good oral hygiene (Full-mouth plaque score <25%).
3. Subject would be available for study monitoring and follow-up visits.
4. Patients with missing teeth in the maxillary posterior region who will require sinus augmentation for implant placement. The patients may be partially or completely edentulous.
5. Patient is a candidate for delayed implant placement approximately 8 months following sinus grafting

Exclusion Criteria:

1. Alcohol, drug dependency.
2. Signs or symptoms of chronic maxillary sinus disease.
3. Current smoker.
4. History of head and neck radiation treatment.
5. Poor health, conditions like uncontrolled diabetes, uncontrolled hypertension or other uncontrolled systemic disease.
6. Physical or psychological reason that might affect the surgical procedure or the subsequent prosthodontic treatment and/or required follow-up examinations.
7. Also, subjects who are nursing or pregnant will be excluded from the study.

Ages: 18 Years to 103 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Lozada, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University school of dentistry, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The unit of enrollment here is one maxillary sinus that qualifies for grafting via lateral window approach. 9 patients were recruited who had 15 qualified maxillary sinus' in this study.
Units Other Than Participants: Sinus augmentation
Period: Overall Study
Arm/Group | InterOss | Bio-oss
Started | 4; 6 Sinus augmentation | 5; 9 Sinus augmentation
Completed | 4; 6 Sinus augmentation | 5; 9 Sinus augmentation
Not Completed | 0; 0 Sinus augmentation | 0; 0 Sinus augmentation

BASELINE CHARACTERISTICS:
Population: These participants were selected for grafting of the maxillary sinus floor based on the minimum availability of the bone present in that area for implant placement.
Units Other Than Participants: Maxillary sinus
Groups:
- Total: Total of all reporting groups
Arm/Group | InterOss | Bio-oss | Total
Number analyzed (Participants) | 4 | 5 | 9
Number analyzed (Maxillary sinus) | 6 | 9 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (4.1) | 54.2 (2.3) | 59.6 (4.3)
Sex: Female, Male [Count of Units; unit: Maxillary sinus] — Population: The unit measured is the number of Maxillary sinus. The participants are number of people in the study. Some of the patients had one maxillary sinus that qualified for the study and some of the patients had both maxillary sinuses that qualified for the study.
  Maxillary sinus
    Female | 3 | 2 | 5
    Male | 3 | 7 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of New Vital Bone.
Description: Vital bone as seen in histology from the collected bone cores.
Time Frame: 8 months post operative after the initial sinus augmentation surgery.
Population: Subjects requiring sinus augmentation for implant placement
Measure: Mean (Standard Deviation); unit: percentage of new vital bone
Units Other Than Participants: Sinus
Arm/Group | InterOss | Bio-oss
Number analyzed (Participants) | 4 | 5
Number analyzed (Sinus) | 6 | 9
percentage of new vital bone
  Lateral core | 16.33 (8.43) | 26.11 (11.63)
  Crestal core | 30.5 (5.86) | 39.67 (3.52)

2. Secondary Outcome: Cumulative Percentage of Bone Marrow and Fibrous Tissue
Description: Cumulative percentage of Bone marrow and fibrous tissue as seen in histology.
Time Frame: Eight months post-op sinus augmentation
Population: Subjects requiring sinus augmentation for implant placement
Measure: Mean (Standard Deviation); unit: Cumulative percentage
Arm/Group | InterOss | Bio-oss
Number analyzed (Participants) | 4 | 5
Cumulative percentage
  Lateral core | 56.33 (5.57) | 51.67 (6.48)
  Crestal core | 50.17 (5.53) | 46.33 (8.91)

3. Secondary Outcome: Space
Description: Space seen the histology specimen not filled with either bone or fibrous tissue in the bone core specimens.
Time Frame: 8 months
Population: Subjects requiring sinus augmentation for implant placement
Measure: Mean (Standard Deviation); unit: percentage of space not filled with bone
Arm/Group | InterOss | Bio-oss
Number analyzed (Participants) | 4 | 5
percentage of space not filled with bone
  Lateral core | 27.33 (13.54) | 22.11 (10.15)
  Crestal core | 19.5 (4.59) | 14.00 (12.51)

ADVERSE EVENTS:
Time Frame: Adverse events data collected through nine months after sinus augmentation
Arm/Group | InterOss | Bio-oss
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT03059914/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT03059914/ICF_001.pdf